CLINICAL TRIAL: NCT02771548
Title: Biomechanical Analysis of Dynamic Tasks and Muscular Strength Following Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Dr Neil Welch ASCC (Other)
Collaborators: Sports Surgery Clinic Research Foundation (Unknown); Insight Centre for Data Analytics (Other); Science Foundation Ireland (Other); University of Roehampton (Other); University of Melbourne (Other); University College Cork (Other); University of Leeds (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Dr Neil Welch ASCC, Head of lab services and research, Sports Surgery Clinic, Santry, Dublin
Organization: Sports Surgery Clinic, Santry, Dublin (Other)
Other Study IDs: SSC-ACL-001
Record Dates: First submitted 2016-02-05; First posted 2016-05-13 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Knee injuries; Rehabilitation; Return to sport; Biomechanics
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (2):
- Anterior Cruciate Ligament Reconstruction: Those who have undergone unilateral anterior cruciate ligament reconstructive surgery in the Sports Surgery Clinic.
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction
- Control: Healthy volunteers with no previous knee injury, no current lower limb injuries and take part in regular multidirectional team sports.

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament Reconstruction
  Groups: Anterior Cruciate Ligament Reconstruction

SUMMARY:
Background

Anterior cruciate ligament (ACL) injuries are one of the most common sporting injuries of the knee. ACL reconstruction (ACLR) has become one of the most common surgical procedures in an attempt to increase joint stability and facilitate athletes to return to sport (RTS). Although ACLR is considered a relatively successful procedure, dynamic control risk factors and strength and power deficits in the involved limb are still present after patients return to sport.

Dynamic multi-plane, multi-joint actions such as jumping, landing, change of direction cutting, have been shown to be common mechanisms of injury for the ACL in field sports . Returning to multidirectional sports requires a proficiency and efficiency of movement when carrying out these tasks. There is a lack of standardized, objective criteria to accurately assess an athlete's ability to safely RTS. Therefore, there is a need for research that simultaneously analyses sport specific dynamic tasks (3D motion analysis) and muscular strength/power deficits that may explain poor outcomes following ACLR. This study aims to further investigate movement patterns, limb asymmetry and muscle strength deficit in patients post-surgery to identify risk factors for re-injury and criteria for RTS.

The purpose of this study was to:

1. Analyse kinematic (movement descriptors) and kinetic (forces that cause movement) during sports specific dynamic tasks at different time-points (6 and 9 months) following ACLR.
2. To explore the association of those findings with those who re-injure, those who have persistent knee pain or with those who fail to return to sport.
3. To compare the ACLR participants with age and gender matched healthy multidirectional athletes.

It is hypothesised that biomechanical analysis will identify clear risk factors for poor outcomes following ACLR. Analysis of ACLR athletes' biomechanics during sports specific tasks will aid in the identification of athletes who are not yet ready to return to sport and will inform the clinician of what must be targeted in specific rehabilitation protocols before return to sport is considered.

Brief protocol

Participants will be recruited from patients who are scheduled to undergo anterior cruciate ligament reconstruction at the Sports Surgery Clinic, Ireland. Healthy participants will be recruited from local multidirectional teams. Participation will be voluntary and after obtaining informed consent patients will be asked to complete pre-operative questionnaires to ascertain injury information, and the function of their knee. During surgery the surgeon will fill out an intra-operative questionnaire. Items recorded will include graft type, laxity, involvement of other ligamentous structures, type of femoral and tibial fixation, meniscal or chondral pathology.

Biomechanical assessment takes place at 6 and 9 months post surgery for the ACL group while the healthy participants will be tested on one occasion. The 3D testing session will include capturing of jumping, landing, hopping and cutting mechanics through the use of three dimensional motion capture technology and force plates. Here reflective markers are placed on the skin at anatomical landmarks. These markers are picked up by the infrared cameras and tracked at 200 frames per second. Participants will make contact with a force plate with their foot on undertaking the movements. Force and marker data will be combined to calculate joint angles and moments. Participants will also perform a muscle strength test using equipment called an isokinetic dynamometer. Both the operated and non-operated limbs will be tested.

Participants will also be asked to fill out validated questionnaires to monitor self reported knee function, their confidence in their knee and also collect data on any continuing adverse symptoms such as locking, giving way, swelling or pain. Participants will also be asked if and when they return to sport. Questionnaires will be administered to participants at pre-op, 3, 6, 9, 12, 24 months, 5 and 10 years post operatively.

DETAILED DESCRIPTION:
3D Biomechanical testing involves the following progressive neuromuscular challenge tests:

* Single leg countermovement jump - Vertical jump as high as possible off one leg.
* Single leg drop jump- Hop from a 20cm height onto one leg and jump as high as possible with as little time spent on the ground
* Double leg drop jump- Hop from a 30cm height onto one leg and jump as high as possible with as little time spent on the ground
* Hurdle hop - Lateral hop over a 15cm hurdle followed by a hop back to the starting position and a hold for 2sec
* Single Leg Hop for distance - maximal jump for horizontal distance on one leg while sticking the landing
* Pre-planned change of direction cut - Sprint for 5 metres, make a 90 degree change of direction pre-determined by the tester and sprint for a further five meters to the finish
* Indecision cut - Sprint for five meters then react to a light stimulus and make a 90 degree cut to the left or right for a further 1.5metres

Patient Registry

Patient data will be inputted into the Sports Surgery Clinic medical data management software. Captured data will include:

1. Patient information - Date of Surgery, Surgeon, Side of ACLR, confirmative Magnetic Resonance Imaging
2. Pre-Operative data collection

   * Pre-Operative Questionnaire- Date of injury, Activity undertaking when injury occurred, level of sporting activity, Injury mechanism, limb dominance, previous ACL injury or surgery.
   * Marx Activity Questionnaire.
   * ACL return to sports after injury (RSI) questionnaire- measures the athlete's emotions, confidence in performance, and risk appraisal in relation to return to sport after an ACL injury.
3. Intra-Op data collection

   - Operative notes are recorded in theatre using a standardised in theatre questionnaire. This form was developed under consensus with all surgeons who complete ACL reconstructive surgery at the Sports Surgery Clinic. Included are graft type, laxity, involvement of other ligamentous structures, type of femoral and tibial fixation, meniscal or chondral pathology.
4. 6 Month and 9 months post op data collection

   * Marx Activity Questionnaire
   * ACL RSI
   * International Knee Documentation Committee (IKDC) form- The IKDC subjective form is a reliable and valid measure to monitor symptoms and function in daily living activities in those with knee disorders.
   * Cincinnati Questionnaire - a valid and reliable measure of patient reported outcome after ACL injury
   * Sports Surgery Clinic return to performance questionnaire- asks whether the participant has returned to sport, have they injured the operated knee or contralateral knee and asks whether they still experience pain and rate that pain on a numerical rating scale.
   * 3D test battery findings
5. 12 and 24 months post op data collection

   * Marx Activity Questionnaire
   * ACL RSI
   * IKDC
   * Sports Surgery Clinic return to performance questionnaire

Quality assurance plan

* Weekly cross-checking will be undertaken by two members of staff to ensure data entered onto the registry is correct and contemporaneous.
* A six-monthly audit of the registry will be undertaken by external auditors.

Registry standard operating procedures

* Basic patient contact details are inputted by administration staff.
* Physiotherapists and biomechanists input physical examination findings on medical data software.
* Self-reported questionnaires are completed on site using a tablet device and uploaded automatically to the registry once the questionnaire is completed.
* During theatre, the surgeon fills out the standardised intra-operative form, which is uploaded to the registry following surgery.
* For analysis or auditing purposes, data is downloaded from the Sports Surgery Clinic medical data management software and placed into Microsoft excel. Patient names are de-identified.

Sample size

* Suggested sample size = 1000
* Sample size calculation was carried out based on current numbers presenting to the clinic. Clinical numbers indicate a re-rupture rate of either the ipsilateral or contralateral ACL of 5%.
* This study aims to recruit 1000 participants and follow them over 24 months. With a likely re-rupture rate of 5%- it is hypothesized that 50 re-ruptures will occur over the 24 month period. This is a conservative number allowing for dropouts, and a split between contralateral and ipsilateral ACL injuries, which will be analysed separately.
* It is also aimed to recruit 50 healthy volunteers from multidirectional field sports teams.

Plan for missing data

* Checklist to flag missing data at the end of every week
* Participants with missing data may be excluded from the data analysis.

Statistical analysis plan

* Variables of interest include kinematics, kinetics, power, and vertical ground-reaction force at the pelvis, hip, knee and ankle at specific time points during different jumping, landing and cutting manoeuvres.
* Differences between involved and uninvolved legs will be calculated, and used to assess for asymmetry. Two group comparisons will be conducted using the Student t test or Kruskal-Wallis test for normal and non-normally distributed variables, respectively.
* Multivariable logistic regression, using variables with P values of </=0.05 from 2-group comparisons (those who go on to suffer a 2nd ACL injury and those who don't), will be used to identify the most predictive variables of the second ACL injury.
* A multivariable logistic regression analysis will also be conducted to identify the most predictive variables of patient reported subjective knee function (IKDC) and pain.
* Associations between intra-operative findings and outcome measures of re-injury pain and return to sport will be explored, also using regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Active participants
* Anterior cruciate ligament reconstruction surgery in the Sports Surgery Clinic.
* Over the age of 13 years

Exclusion Criteria:

* Multiple orthopaedic injuries concurrently.
* Surgery outside of Sports Surgery Clinic.

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Those who undergo anterior cruciate ligament reconstruction in the Sports Surgery Clinic, Dublin, and who meet the inclusion criteria, will be asked if they wish to participate in this study. Sports Surgery Clinic is a private hospital where over 750 ACL reconstructive surgeries take place each year. Many patients will travel from all over the country of Ireland to the clinic for the surgery, meaning there is a wide catchment area for participants.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Return to Performance- change in status | 6,9,12 and 24 months post operatively
  The Sports Surgery Clinic return to performance questionnaire asks whether the participant has returned to sport.
Injured operated knee- change in status | 6,9,12 and 24 months post operatively
  Participants are asked have they injured their operated knee.
Injured their contralateral knee- change in status | 6,9,12 and 24 months post operatively
  Participants are asked have they injured their operated knee.
Change in pain experienced | 6,9,12 and 24 months post operatively
  Participants will be asked to rate their pain on a numerical rating scale, 0-10.

SECONDARY OUTCOMES:
Change in Kinetic and kinematic composite score of the lower limb, pelvis and trunk | At 6 and 9 months post surgery
  Associations can be made between post surgical change in biomechanical variables exhibited on sports specific tasks and poor outcomes following ACLR.
Change in International Knee Documentation Committee (IKDC) | 3, 6, 9, 12 and 24 months post surgery
  The IKDC subjective form is a reliable and valid measure to monitor symptoms and function in daily living activities in those with knee disorders (Higgins et al. 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Ray Moran, MCh (Orth) FRCSI FFSEM, Study Director — Sports Surgery Clinic; Mark Jackson, MBBS BSc FRCS, Study Director — Sports Surgery Clinic
Locations (1):
- Sports Surgery Clinic, Dublin, Leinster, Ireland

REFERENCES:
- [Background] Boden BP, Griffin LY, Garrett WE Jr. Etiology and Prevention of Noncontact ACL Injury. Phys Sportsmed. 2000 Apr;28(4):53-60. doi: 10.3810/psm.2000.04.841. PMID 20086634
- [Background] Koga H, Nakamae A, Shima Y, Iwasa J, Myklebust G, Engebretsen L, Bahr R, Krosshaug T. Mechanisms for noncontact anterior cruciate ligament injuries: knee joint kinematics in 10 injury situations from female team handball and basketball. Am J Sports Med. 2010 Nov;38(11):2218-25. doi: 10.1177/0363546510373570. Epub 2010 Jul 1. PMID 20595545
- [Background] Higgins LD, Taylor MK, Park D, Ghodadra N, Marchant M, Pietrobon R, Cook C; International Knee Documentation Committee. Reliability and validity of the International Knee Documentation Committee (IKDC) Subjective Knee Form. Joint Bone Spine. 2007 Dec;74(6):594-9. doi: 10.1016/j.jbspin.2007.01.036. Epub 2007 Aug 6. PMID 17888709
- [Background] Marx RG, Stump TJ, Jones EC, Wickiewicz TL, Warren RF. Development and evaluation of an activity rating scale for disorders of the knee. Am J Sports Med. 2001 Mar-Apr;29(2):213-8. doi: 10.1177/03635465010290021601. PMID 11292048
- [Background] Webster KE, Feller JA, Lambros C. Development and preliminary validation of a scale to measure the psychological impact of returning to sport following anterior cruciate ligament reconstruction surgery. Phys Ther Sport. 2008 Feb;9(1):9-15. doi: 10.1016/j.ptsp.2007.09.003. Epub 2007 Nov 5. PMID 19083699
- [Background] Barber-Westin SD, Noyes FR, McCloskey JW. Rigorous statistical reliability, validity, and responsiveness testing of the Cincinnati knee rating system in 350 subjects with uninjured, injured, or anterior cruciate ligament-reconstructed knees. Am J Sports Med. 1999 Jul-Aug;27(4):402-16. doi: 10.1177/03635465990270040201. PMID 10424208
- [Background] Paterno MV, Schmitt LC, Ford KR, Rauh MJ, Myer GD, Huang B, Hewett TE. Biomechanical measures during landing and postural stability predict second anterior cruciate ligament injury after anterior cruciate ligament reconstruction and return to sport. Am J Sports Med. 2010 Oct;38(10):1968-78. doi: 10.1177/0363546510376053. Epub 2010 Aug 11. PMID 20702858
- [Derived] McAleese T, Welch N, King E, Roshan D, Keane N, Moran KA, Jackson M, Withers D, Moran R, Devitt BM. Primary Anterior Cruciate Ligament Reconstruction in Level 1 Athletes: Factors Associated With Return to Play, Reinjury, and Knee Function at 5 Years of Follow-up. Am J Sports Med. 2025 Mar;53(4):777-790. doi: 10.1177/03635465241313386. Epub 2025 Feb 7. PMID 39919304
- [Derived] King E, Richter C, Daniels KAJ, Franklyn-Miller A, Falvey E, Myer GD, Jackson M, Moran R, Strike S. Biomechanical but Not Strength or Performance Measures Differentiate Male Athletes Who Experience ACL Reinjury on Return to Level 1 Sports. Am J Sports Med. 2021 Mar;49(4):918-927. doi: 10.1177/0363546520988018. Epub 2021 Feb 22. PMID 33617291
- [Derived] King E, Richter C, Daniels KAJ, Franklyn-Miller A, Falvey E, Myer GD, Jackson M, Moran R, Strike S. Can Biomechanical Testing After Anterior Cruciate Ligament Reconstruction Identify Athletes at Risk for Subsequent ACL Injury to the Contralateral Uninjured Limb? Am J Sports Med. 2021 Mar;49(3):609-619. doi: 10.1177/0363546520985283. Epub 2021 Feb 9. PMID 33560866
- [Derived] King E, Richter C, Jackson M, Franklyn-Miller A, Falvey E, Myer GD, Strike S, Withers D, Moran R. Factors Influencing Return to Play and Second Anterior Cruciate Ligament Injury Rates in Level 1 Athletes After Primary Anterior Cruciate Ligament Reconstruction: 2-Year Follow-up on 1432 Reconstructions at a Single Center. Am J Sports Med. 2020 Mar;48(4):812-824. doi: 10.1177/0363546519900170. Epub 2020 Feb 7. PMID 32031870
- [Derived] King E, Richter C, Franklyn-Miller A, Wadey R, Moran R, Strike S. Back to Normal Symmetry? Biomechanical Variables Remain More Asymmetrical Than Normal During Jump and Change-of-Direction Testing 9 Months After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2019 Apr;47(5):1175-1185. doi: 10.1177/0363546519830656. PMID 30943079